CLINICAL TRIAL: NCT04593875
Title: Low-Intensity Focused Ultrasound Pulsation for Treatment of Motor Deficits in Parkinson's Disease
Brief Title: LIFUP for Treatment of Motor Deficits in Parkinson's Disease
Acronym: LIFUP PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Susan Bookheimer, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#20-001901
Record Dates: First submitted 2020-10-03; First posted 2020-10-20 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: LIFUP; Ultrasound
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to both study arms; the order in which they complete the arms will be randomized and counterbalanced. The two visits will be spaced apart by 2 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants complete two identical in-person testing and LIFUP sessions. At one session, the device will be used with a gel pad that allows ultrasound to pass through, and at the other session, it will be used with a gel pad that blocks the ultrasound. The order of conditions is randomized and counterbalanced across participants. The two gel pads look identical beyond a label differentiating them, and neither the participants nor the person administering ultrasound will know whether sham or active is being administered at a given session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active, then Sham (Experimental): Active Low intensity focused ultrasound pulsation (LIFUP) will be administered to the internal globus pallidus while participants are in the MRI scanner. Then, 2 weeks later, sham LIFUP will be administered.
  Interventions: Device: Active LIFUP Treatment; Device: Sham LIFUP Treatment
- Sham, then Active (Experimental): Sham low intensity focused ultrasound pulsation (LIFUP) will be administered while participants are in the MRI scanner. Then, 2 weeks later, active LIFUP will be administered to the internal globus pallidus.
  Interventions: Device: Active LIFUP Treatment; Device: Sham LIFUP Treatment

INTERVENTIONS:
Device: Active LIFUP Treatment — Low intensity focused ultrasound pulsation will be administered to the internal globus pallidus in 20 sonications at 650kHz, ispta.3 720mW/cm, pulse repetition frequency 100Hz, duty cycle 5%, duration 30s with 30s spacing between sonications. For active LIFUP, the device will be used with a gel pad that allows the ultrasound to pass through.
  Other Names: BX Pulsar 1002
Device: Sham LIFUP Treatment — The device will be aimed at the internal globus pallidus and turned on with the same settings as the active condition; however, in this case, the device will be used with a gel pad that blocks the ultrasound from passing through, such that no ultrasound is actually being administered to the brain.

SUMMARY:
The study will test the feasibility of using Low Intensity Focused Ultrasound Pulsation (LIFUP) to treat motor symptoms in Parkinson's Disease (PD). LIFUP is a new technique that can increase brain activity in highly specific target areas and is MRI compatible. Thus, in real-time, it is possible to directly observe how LIFUP changes the brain areas important in PD by measuring its effects on brain activity, blood flow, and brain connectivity. If successful, this research will mark the first step towards a novel, non-invasive, non-medication treatment for PD.

DETAILED DESCRIPTION:
This trial is a proof-of-concept, proof-of-mechanism study of a novel neuromodulation technology - LIFUP - to treat motor symptoms in PD. Much like Deep Brain Stimulation, LIFUP can be focused on deep brain structures with high spatial accuracy, including those implicated in PD; however, it can do so non-invasively. Other non-invasive neuromodulation tools such as Transcranial Magnetic Stimulation can only target surface brain structures and are not optimal PD treatment tools. This study will test this new technology in 30 participants with PD during simultaneous resting state functional MRI, and collect pre- and post-LIFUP functional MRI, arterial spin labeling, motor performance data, and behavioral data, in a double-blind crossover trial to determine whether LIFUP: 1) will improve motor symptoms during and after treatment; 2) can modulate neural activity in the target brain region important for PD, the internal globus pallidus; and 3) enhance cortico-striatal motor circuit connectivity. All participants in this study will receive active ultrasound at one of the two in-person sessions and sham at the other.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Age 18-85
3. Fluent in the English language

Exclusion Criteria:

1. Metal implants that are not MR compatible
2. Neurological diagnosis other than Parkinson's
3. Not fluent in the English language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Y Bookheimer, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (1 day)
Arm/Group | Active, Then Sham | Sham, Then Active
Started | 15 | 16
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Washout / Follow-Up (2 weeks)
Arm/Group | Active, Then Sham | Sham, Then Active
Started | 15 | 16
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Withdrawn by investigator after completing first intervention follow-up | 0 | 1
Period: Second Intervention (1 day)
Arm/Group | Active, Then Sham | Sham, Then Active
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention Follow-Up (1 week)
Arm/Group | Active, Then Sham | Sham, Then Active
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant in the "sham then active" group was withdrawn after their first in-person session due to excessive head motion in the MRI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active, Then Sham | Sham, Then Active | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.5) | 66.8 (8.0) | 66.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 16 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Motor Assessment 1: Unified Parkinson Disease Rating Scale (UPDRS) Section 3
Description: The participant will complete a 18-item comprehensive motor assessment that assesses elements of motor function including tremor, bradykinesia, and gait. The total score for this assessment ranges from 0 to 108 points, with higher scores indicating higher severity.
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: One participant was not included in motor symptom analyses due to extreme motor symptom fluctuations at baseline confounding measurement of LIFUP-related changes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active LIFUP Session: LIFUP will be administered to the internal globus pallidus on the side of the brain contralateral to the side of the body with worse symptoms. The side of the brain contralateral to worse symptoms is being targeted because the left hemisphere of the brain primarily controls right side motor function and vice versa.
  The LIFUP protocol will entail 20 sonications at 650kHz, 720mW/cm, duty cycle 5%, pulse repetition frequency 100Hz, duration 30s, with 30s spacing between sonications.
- Sham LIFUP Session: LIFUP will be administered with an identical protocol to the active session; however, the gel pad used during the sham session blocks the ultrasound such that none actually reaches the head.
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 29 | 29
score on a scale
  Pre-LIFUP | 37.24 (9.91) | 35.14 (8.28)
  Post-LIFUP | 36.93 (9.54) | 34.21 (9.43)

2. Primary Outcome: Motor Assessment 2: Finger Tapping (Score)
Description: This task, which is item 3.4 on the Unified Parkinson's Disease Rating Scale (UPDRS), asks participants to tap their index finger on their thumb ten times as big and as fast as possible. Participants scores on item 3.4 with standard UPDRS scoring criteria (on a scale of 0 to 4, where a higher score indicates more severe Parkinson's symptoms i.e. worse performance) will be assessed pre and post-LIFUP. The scores reported below are for the hand on the side with worse symptoms (i.e. the side that LIFUP is intended to primarily affect).
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 29 | 29
score on a scale
  Pre-LIFUP Score | 1.48 (0.829) | 1.45 (0.936)
  Post-LIFUP Score | 1.66 (0.974) | 1.34 (0.948)

3. Primary Outcome: Motor Assessment 2: Finger Tapping (Speed)
Description: This task, which is item 3.4 on the Unified Parkinson's Disease Rating Scale (UPDRS), asks participants to tap their index finger on their thumb ten times as big and as fast as possible. The speed of taps will be assessed pre and post-LIFUP. Speed is calculated as [number of taps per second] times [average tap amplitude], where tap amplitude is measured on a scale of 0.0-1.0 representing the percentage of finger extension between taps, where e.g. extension to a 90 degree angle between thumb and index finger = 1.0, extension to 45 degree angle = 0.5, etc. Higher speed indicates better performance. The speed values reported below are for the hand on the side with worse symptoms (i.e. the side that LIFUP is intended to primarily affect).
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Measure: Mean (Standard Deviation); unit: tap amplitude per second
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 29 | 29
tap amplitude per second
  Pre-LIFUP Speed | 1.81 (0.75) | 1.72 (0.74)
  Post-LIFUP Speed | 1.70 (0.75) | 1.94 (0.80)

4. Primary Outcome: Motor Assessment 2: 9-Hole Pegboard Dexterity Test
Description: The participant will place and remove nine plastic pegs into a plastic pegboard. Scores are recorded as time in seconds that it takes the participant to complete the task with each hand. Analysis will compare pre- and post-treatment scores to quantify motor performance improvements.
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 29 | 29
Seconds
  Pre-LIFUP (Hand on side with more severe symptoms) | 23.87 (9.44) | 23.94 (9.61)
  Post-LIFUP (Hand on side with more severe symptoms) | 23.49 (7.54) | 23.12 (7.34)
  Pre-LIFUP (Hand on side with less severe symptoms) | 21.04 (6.26) | 20.73 (7.50)
  Post-LIFUP (Hand on side with less severe symptoms) | 20.46 (5.79) | 20.12 (4.40)

5. Secondary Outcome: Difference in BOLD fMRI Signal Between on vs. Off Blocks
Description: BOLD data will be collected in real-time during the ultrasound sonication, which occurs in interleaved 30 second "on" and "off" blocks. Analyses will assess the statistical relationship between BOLD signal in the brain and the time series (on vs off) of the ultrasound sonication. Tabular data reported here represents the difference in BOLD activation between on and off conditions in the internal globus pallidus on the targeted side of the brain, calculated as the mean BOLD activation while LIFUP is on minus mean activation when it is off.
Time Frame: During LIFUP (or sham) sonication on Day 1 and Day 15
Population: Three participants were excluded from this analysis due to excessive motion or preprocessing failure.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 27 | 27
BOLD signal change | 1.19 (6.53) | 0.41 (3.49)

6. Secondary Outcome: Perfusion Changes in Internal Globus Pallidus, External Globus Pallidus, and Putamen
Description: Arterial spin labeling data will be collected before and after sonication. Analyses will assess the statistical relationship between perfusion in the targeted internal globus pallidus, external globus pallidus, and putamen pre- and post-sonication in a within-subject repeated measures design.
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: Data from the active session from 11 participants and from the sham session for 5 participants were excluded due to incomplete data or image reconstruction or preprocessing failures.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active LIFUP Session | Sham LIFUP Session
Number analyzed (Participants) | 19 | 25
percentage change
  GPi - Percent Change Perfusion | 16.4 (50.6) | 17.0 (50.1)
  GPe - Percent Change Perfusion | 30.0 (101.2) | 16.6 (46.1)
  Putamen - Percent Change Perfusion | 28.4 (63.4) | 14.0 (45.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 2, 4, and 7 days after each in-person session, and the two in-person sessions were two weeks apart. As a result, depending on whether participants received active then sham or sham then active, adverse event data were collected for either one week or three weeks after the active intervention.
Description: Participants were asked a series of open-ended questions 2, 4, and 7 days after each in-person sessions, as well as at the start of their second in person session (i.e. 2 weeks after session 1) . These questions asked participants if they had observed any 1. changes in impulsivity, anxiety, mood, or thinking skills, 2. motor changes, and 3. other changes, as well as if they had any other comments.
Arm/Group | Active LIFUP Session | Sham LIFUP Session
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 5/30 | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active LIFUP Session (N=30) | Sham LIFUP Session (N=31)
Head or Neck Pain (Nervous system disorders) | 2 | 3 — Participants reporting headache, neck pain, or local pain on scalp at site of device during or after LIFUP or sham procedure
Fatigue or Sleep Disruption (General disorders) | 3 | 3 — Self-reported fatigue or other alterations to sleep patterns (insomnia, excessive sleep)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04593875/Prot_SAP_000.pdf